CLINICAL TRIAL: NCT04895488
Title: Cognitive Effects of Adjuvant Vortioxetine in Early Schizophrenia
Acronym: CAVES
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAVES; 2021-001333-38 (EudraCT Number)
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Impairment With Primary Psychotic Disorder; Negative Symptoms With Primary Psychotic Disorder
MeSH Terms: interventions — Vortioxetine

STUDY DESIGN:
Intervention Model Description: A two arm, Open-label, randomized, Cross-over Design and single-center clinical trial Phase II b /Phase III.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Vortioxetine+Usual antipsychotic treatment (TAU) (Experimental): Drug:
  First treatment phase: Vortioxetine 10 mg 1 tablet/d for 2 weeks added to Usual antipsychotic treatment, followed by Vortioxetine 20mg 1tablet/d for 22 weeks added to Usual antipsychotic treatment.
  Wash-out period 2 weeks
  Interventions: Drug: Vortioxetine; Drug: Usual Antipsychotic Treatment
- Arm B: Usual antipsychotic treatment (TAU) (Active Comparator): Second treatment phase: Usual antipsychotic treatment: Allows for whatever medication, routine support, or referral to other services was felt appropriate by the clinician.
  Interventions: Drug: Vortioxetine; Drug: Usual Antipsychotic Treatment

INTERVENTIONS:
Drug: Vortioxetine — First treatment phase: vortioxetine will be initiated at 10 mg / day for 2 weeks, followed by 20 mg /day for 22 weeks. The dose of vortioxetine can be lowered to 5 mg or 10 mg for tolerability reasons at clinician criteria.
  Wash-out period 2 weeks
Drug: Usual Antipsychotic Treatment — Second treatment phase. Usual antipsychotic treatment for 26 weeks: Allows for whatever medication, routine support, or referral to other services was felt appropriate by the clinician.
  Other Names: TAU

SUMMARY:
Clinical trial to assess the efficacy of Vortioxetine compared with treatment as usual in early schizophrenia.

DETAILED DESCRIPTION:
Clinical trial to assess the efficacy of Vortioxetine, compared with treatment as usual in early schizophrenia. Propose: To investigate the effect of Vortioxetine in cognitive functioning and negative symptoms severity in early schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient
2. Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders (DSM - SCID) diagnosis of Schizophrenia spectrum disorders.
3. Age >18-50 years old
4. Stable antipsychotic medication doses during at least 4 weeks ( all second generation antipsychotics excluding clozapine).
5. No antidepressant treatment for at least 8 weeks prior to randomization.
6. PANSS Negative subscore >14 with at least two of the items at a level >/=4 (moderate)
7. PANSS Positive subscore </=14 with not more than one of the items at a level >/=4 (moderate)
8. Hamilton Depression Rating Scale (HAMD-17) total score </=12
9. Simpson Angus Score of any item <2
10. Behaviorally Anchored Rating Scale (BARS) of any item </= 1
11. Competent and willing to sign informed consent
12. The patient, if a woman, must: agree not to try to become pregnant during the study and use adequate, highly effective contraception

Exclusion Criteria:

1. Patients taking any antidepressant and its use cannot be discontinued at least 8 weeks prior to randomization.
2. Structural brain disease (based on previous medical records)
3. Cognitive disability by history and estimated intelligence quotient (IQ) <70 (ID DSM-5 diagnosis).
4. Any serious chronic medical illnesses that may interfere with the patient's ability to comply with the study procedures or that will interfere with cognition.
5. Organic mental disorders, or mental disorders due to a general medical condition. Any neurological or neurodegenerative disorders.
6. Any current diagnosis of substance abuse or dependence.
7. Serious risk of suicide.
8. Patients with thyroid conditions.
9. Intolerance to or inefficacy of vortioxetine in the past. Patients who had failed treatment with vortioxetine were also excluded.
10. Pregnant or breastfeeding female.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of Vortioxetine vs. TAU measured by the change in Brief Assessment of Cognition in Schizophrenia (BACS App) scores | Baseline, week 24, week 26 and week 50
  To assess the effectiveness of Vortioxetine vs. TAU in the treatment of cognitive impairments in early psychosis, measured by the change From Baseline to Week 24 in BACS App scores using the Composite Z-score Defined as the Weighted Sum of the Individual Patient Z-scores

SECONDARY OUTCOMES:
To assess the effectiveness of Vortioxetine vs. TAU measured by the change in Negative Symptoms severity (Scale for Assessment of Negative Symptoms (SANS) and Negative Symptom Assessment-4 (NSA-4) total scores) | Baseline, week 4, week 12, week 24, week 26, week 30, week 38 and week 50
  To assess the effectiveness of Vortioxetine vs. TAU in the treatment of negative symptoms in early psychosis, measured by the change in Negative Symptoms severity (SANS, NSA-4 total scores) from baseline to end of trial.

OTHER OUTCOMES:
To assess the effectiveness of Vortioxetine vs. TAU measured by the change in general functioning | baseline, week 12, week 24, week 26, week 38 and week 50
  To assess the effectiveness of Vortioxetine vs. TAU in the treatment of cognitive impairments in early psychosis, measured by the change in general functioning (Global Assessment of Functioning (GAF) total score)
To assess the safety of Vortioxetine measured through the communication of any serious adverse event. | from informed consent form (ICF) signature to 52 weeks
  To assess the safety of Vortioxetine in patients with early psychosis measured through the communication of any serious adverse event evaluated for relationship with the Investigational Medicinal Product (IMP).

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo Facorro, Professor, Principal Investigator — benedicto.crespo.sspa@juntadeandalucia.es
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

DOCUMENTS (1):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT04895488/Prot_000.pdf